CLINICAL TRIAL: NCT07027293
Title: Evaluation of the Insertion of I-gel and Classic LMA in Different Head Positions in Elderly Patients
Brief Title: The Insertion of I-gel and Classic LMA in Different Head Positions in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Yadigar Yılmaz, MD, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: E-10840098-202.3.02-1265
Record Dates: First submitted 2025-05-27; First posted 2025-06-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Airway Management Assessment; Supraglottic Airways; Supraglottic Airways for General Anesthesia; Laryngeal Mask Airways
Keywords: Supraglottic airway device; i-gel; Classic laryngeal mask airway; Elderly patients; Airway management; Head position; General anesthesia; Insertion success

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard head position + i-gel (Active Comparator)
  Interventions: Other: STANDART HEAD POSITION; Device: i-gel supraglottic airway device
- Rotated head position + i-gel (Active Comparator)
  Interventions: Other: HEAD ROTATION POSITION; Device: i-gel supraglottic airway device
- Standard head position + classic LMA (Active Comparator)
  Interventions: Other: STANDART HEAD POSITION; Device: Classic laryngeal mask airway (LMA)
- Rotated head position + classic LMA (Active Comparator)
  Interventions: Other: HEAD ROTATION POSITION; Device: Classic laryngeal mask airway (LMA)

INTERVENTIONS:
Other: STANDART HEAD POSITION — STANDART HEAD POSITION
  Arms: Standard head position + classic LMA; Standard head position + i-gel
Other: HEAD ROTATION POSITION — HEAD ROTATION POSITION
  Arms: Rotated head position + classic LMA; Rotated head position + i-gel
Device: Classic laryngeal mask airway (LMA) — Classic laryngeal mask airway (LMA)
  Arms: Rotated head position + classic LMA; Standard head position + classic LMA
Device: i-gel supraglottic airway device — i-gel supraglottic airway device
  Arms: Rotated head position + i-gel; Standard head position + i-gel

SUMMARY:
This prospective, randomized, double-blind clinical study aims to evaluate the insertion success of two supraglottic airway devices, the classic Laryngeal Mask Airway (LMA) and the I-gel, in different head and neck positions in elderly patients undergoing elective urological surgery under general anesthesia. A total of 120 patients aged over 75 years with ASA physical status I-III will be randomly assigned to one of four groups: standard position with I-gel, right lateral rotation with I-gel, standard position with classic LMA, and right lateral rotation with classic LMA. The study will compare insertion time, ease and success of placement, number of attempts, hemodynamic responses, oropharyngeal leak pressures, fiberoptic scores, and airway-related complications. The findings aim to provide clinical guidance on the optimal use of supraglottic airway devices in geriatric patients in various head positions.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I-III
* Age over 75 years

Exclusion Criteria:

* Known or anticipated difficult airway
* Contraindications for the use of a supraglottic airway device
* Patients scheduled for endotracheal intubation

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Insertion Time of Supraglottic Airway Device | 1-10 minutes
Number of attempts for LMA replacement | 15-200 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Yadigar Yılmaz, Istanbul, Turkey (Türkiye)